CLINICAL TRIAL: NCT06141486
Title: A Randomized, Double-blind, Phase 3 Study Comparing Efficacy and Safety of Frexalimab (SAR441344) to Placebo in Adult Participants With Nonrelapsing Secondary Progressive Multiple Sclerosis
Brief Title: Efficacy and Safety Study of Frexalimab (SAR441344) in Adults With Nonrelapsing Secondary Progressive Multiple Sclerosis
Acronym: FREVIVA
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EFC17504; U1111-1280-7114 (Registry Identifier: ICTRP); 2023-504359-29 (Registry Identifier: CTIS)
Record Dates: First submitted 2023-11-09; First posted 2023-11-21 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Frexalimab (Experimental): Frexalimab IV administration
  Interventions: Drug: Frexalimab; Drug: MRI contrast-enhancing agents
- Placebo (Placebo Comparator): Matching placebo
  Interventions: Drug: Placebo; Drug: MRI contrast-enhancing agents

INTERVENTIONS:
Drug: Frexalimab — SAR441344 Solution for IV infusion
  Arms: Frexalimab
Drug: Placebo — Solution for IV infusion
  Arms: Placebo
Drug: MRI contrast-enhancing agents — IV, as per respective label

SUMMARY:
The purpose of this randomized, double-blind, placebo-controlled, parallel group study is to determine the efficacy of frexalimab in delaying the disability progression and the safety up to 36 months double-blind administration of study intervention compared to placebo in male and female participants with nrSPMS (aged 18 to 60 years at the time of enrollment). People diagnosed with nrSPMS are eligible for enrollment as long as they meet all the inclusion criteria and none of the exclusion criteria. Study details include:

* This event-driven study will end when the target number of 6-month cCDP events is achieved, and the study is expected to last 43 months from randomization of the first participant to the common study end.
* The number of scheduled visits will be up to 25 (including 3 follow-up visits) with a visit frequency of every month for the first 6 months and then every 3 months.
* If the prespecified number of events for 6-month cCDP is not reached by V21/W180, scheduled visits will continue every 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Participant must have a previous diagnosis of RRMS in accordance with the 2017 revised McDonald criteria.
* Participant must have a current diagnosis of SPMS in accordance with the clinical course criteria revised in 2013 endorsed by an Adjudication Committee.
* Participant must have documented evidence of disability progression observed during the 12 months before screening. Eligibility will be analyzed by an Adjudication Committee.
* Absence of clinical relapses for at least 24 months.
* The participant must have an EDSS score at screening from 3.0 to 6.5 points, inclusive.
* Contraceptive use by men and women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.
* For patients eligible to be treated with siponimod: 1) does not tolerate it due to side effects or safety reasons, or 2) has failed siponimod treatment due to perceived lack of efficacy, or 3) has declined siponimod treatment.

Exclusion Criteria:

* The participant has a history of infection or may be at risk for infection.
* The presence of psychiatric disturbance or substance abuse.
* History, clinical evidence, suspicion or significant risk for thromboembolic events, as well as myocardial infarction, stroke, and/or antiphosholipid syndrome and any participants requiring antithrombotic treatment.
* Current hypogammaglobulinemia defined by immunoglobulin levels (IgG and/or IgM) below the lower limits of normal (LLN) at Screening or a history of primary hypogammaglobulinemia. Patients with a history of secondary hypogammaglobulinemia induced by anti-C20 monoclonal antibodies (eg, ocrelizumab, ofatumumab, ublituximab, rituximab) may be considered for study inclusion provided their immunoglobulin levels are within the normal limits (WNL) at time of Screening.
* A history or presence of disease that can mimic MS symptoms, such as, but not limited to neuromyelitis optica spectrum disorder, systemic lupus erythematosus, Sjogren's syndrome, acute disseminated encephalomyelitis, and myasthenia gravis.
* The participant has sensitivity to any of the study interventions, or components thereof, or has a drug or other allergy that, in the opinion of the Investigator, contraindicates participation in the study.
* The participant was previously exposed to frexalimab.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 900 (Estimated)
Dates: Start 2023-12-27 (Actual); Primary Completion 2026-12-23 (Estimated); Study Completion 2028-03-24 (Estimated)

PRIMARY OUTCOMES:
Time to onset of composite confirmed disability progression (cCDP) confirmed over 6 months in the double-blind treatment period | Up to 36 months
  Defined as Increase from the baseline expanded disability status scale (EDSS) score of ≥1.0 point when the baseline is <5.5, or ≥0.5 point when the baseline is ≥5.5, OR Increase of ≥20% from the baseline time in the 9 hole peg test (9HPT),OR Increase of ≥20% from the baseline time in the timed 25 foot walk (T25FW) test

SECONDARY OUTCOMES:
Time to onset of composite cCDP confirmed over 3 months in the double-blind treatment period | Up to 36 months
Time to onset of individual components of the composite, confirmed over 3-months or 6 months in the double-blind treatment period | Up to 36 months
  increase from the baseline EDSS score of ≥1.0 point when the baseline is <5.5, or ≥0.5 point when the baseline is ≥5.5
Time to onset of confirmed disability improvement (CDI) in the double-blind treatment period | Up to 36 months
  defined as decrease from the baseline EDSS score of ≥1.0 or ≥ 0.5 points when baseline is ≤5.5 or >5.5 points, respectively, confirmed over 6 months.
Number of new and/or enlarging T2hyperintense lesions per scan as detected by MRI, and number of new and/or enlarging T2-hyperintense lesions per scan as detected by MRI | Up to 36 months
  defined as the sum of the individual number of new and/or enlarging T2-hyperintense lesions at all scheduled visits starting after baseline up to the end of double-blind treatment period
Percent change in brain volume loss as detected by MRI scans at the end of double-blind treatment period compared to Month 6 | Up to 36 months
Change in cognitive function at the end of double-blind treatment period compared to baseline as assessed by symbol digit modalities test (SDMT) | Baseline, Up to 36 months
Change from baseline in multiple sclerosis impact scale 29 version 2 (MSIS-29v2) questionnaire scores over time in the double-blind treatment period | Baseline, Up to 36 months
Change from baseline in patient reported outcome measurement information system (PROMIS) Fatigue multiple sclerosis (MS)-8a over time in the double-blind treatment period | Baseline, Up to 36 months
Annualized relapse rate during the double-blind treatment period assessed by protocol defined adjudicated relapses | Up to 36 months
Number of participants with adverse events, SAEs, AEs leading to permanent study intervention discontinuation and AE of special interests (AESIs) | Up to 36 months
Number of participants with potentially clinically significant abnormalities (PCSAs) in laboratory tests, ECG, and vital signs during the study period | Up to 36 months
  12-lead ECG (electrocardiogram) will be obtained using an ECG machine that automatically calculates the heart rate and measures PR, QRS, QT, and QTc intervals.
Number of participants with antibody over time | Up to 36 months
Change from baseline in serum Ig levels over time | Up to 36 months
Change from baseline in plasma neurofilament light chain (NfL) levels over time in the double-blind treatment period | Up to 36 months
Frexalimab plasma concentration over time in the double-blind treatment period | Up to 36 months

CONTACTS AND LOCATIONS:
Locations (339):
- United States (103):
  - Alabama Neurology Associates- Site Number : 8400115, Homewood, Alabama
  - St. Joseph's Hospital and Medical Center- Site Number : 8400139, Phoenix, Arizona
  - Honor Health Scottsdale Osborn Medical Center- Site Number : 8400074, Scottsdale, Arizona
  - Perseverance Research Center- Site Number : 8400138, Scottsdale, Arizona
  - Imaging Endpoints- Site Number : 8400050, Scottsdale, Arizona
  - Sutter East Bay Medical Foundation - Berkeley- Site Number : 8400134, Berkeley, California
  - The Neurology Center of Southern California - Carlsbad- Site Number : 8400023, Carlsbad, California
  - University of California Irvine - School of Medicine- Site Number : 8400143, Irvine, California
  - University of California San Diego - La Jolla- Site Number : 8400095, La Jolla, California
  - Kaiser Permanente - Los Angeles Medical Center- Site Number : 8400184, Los Angeles, California
  - University of Southern California, Los Angeles- Site Number : 8400118, Los Angeles, California
  - Hoag Memorial Hospital Presbyterian- Site Number : 8400031, Newport Beach, California
  - Stanford Neuroscience Health Center- Site Number : 8400120, Palo Alto, California
  - Private Practice - Dr. Regina Berkovich- Site Number : 8400005, West Hollywood, California
  - University of Colorado - Anschutz Medical Campus- Site Number : 8400001, Aurora, Colorado
  - Advanced Neurology of Colorado- Site Number : 8400148, Fort Collins, Colorado
  - Yale University School of Medicine- Site Number : 8400081, New Haven, Connecticut
  - Hartford Healthcare Medical Group- Site Number : 8400069, Norwich, Connecticut
  - New England Institute for Clinical Research- Site Number : 8400114, Stamford, Connecticut
  - MedStar Georgetown University Hospital- Site Number : 8400044, Washington D.C., District of Columbia
  - Neurology of Central Florida- Site Number : 8400147, Altamonte Springs, Florida
  - First Choice Neurology - Espinosa Neuroscience Institute- Site Number : 8400169, Boca Raton, Florida
  - MS & Neuromuscular Center of Excellence- Site Number : 8400015, Clearwater, Florida
  - Beth Israel Deaconess Medical Center - Fort Myers- Site Number : 8400041, Fort Myers, Florida
  - Norman Fixel Institute for Neurological Diseases (FIND)- Site Number : 8400054, Gainesville, Florida
  - Mayo Clinic in Florida- Site Number : 8400093, Jacksonville, Florida
  - Neurology Associates - Maitland- Site Number : 8400010, Maitland, Florida
  - University of Miami Hospital- Site Number : 8400177, Miami, Florida
  - Orlando Health Neuroscience Institute - Downtown Pavilion- Site Number : 8400060, Orlando, Florida
  - Axiom Clinical Research of Florida- Site Number : 8400049, Tampa, Florida
  - University of South Florida- Site Number : 8400013, Tampa, Florida
  - Palm Beach Neurology- Site Number : 8400105, West Palm Beach, Florida
  - Velocity Clinical Research - Savannah Neurology- Site Number : 8400061, Savannah, Georgia
  - Joi Life Wellness Group LLC- Site Number : 8400192, Smyrna, Georgia
  - Rush University Medical Center- Site Number : 8400102, Chicago, Illinois
  - University of Chicago Medical Center- Site Number : 8400055, Chicago, Illinois
  - Consultants in Neurology- Site Number : 8400020, Northbrook, Illinois
  - Springfield Clinic 1st - 900 Building- Site Number : 8400043, Springfield, Illinois
  - Neuroscience Institute Center- Site Number : 8400053, Merrillville, Indiana
  - University of Iowa- Site Number : 8400029, Iowa City, Iowa
  - University of Kansas Medical Center- Site Number : 8400084, Kansas City, Kansas
  - College Park Family Care Center - Specialty Center- Site Number : 8400032, Overland Park, Kansas
  - Baptist Health Lexington- Site Number : 8400149, Lexington, Kentucky
  - NeuroMedical Clinic of Central Louisiana- Site Number : 8400159, Alexandria, Louisiana
  - The NeuroMedical Center- Site Number : 8400182, Baton Rouge, Louisiana
  - Ochsner Medical Center - Jefferson Highway- Site Number : 8400027, New Orleans, Louisiana
  - University of Maryland School of Medicine - Baltimore- Site Number : 8400185, Baltimore, Maryland
  - Johns Hopkins Hospital- Site Number : 8400080, Baltimore, Maryland
  - International Neurorehabilitation Institute- Site Number : 8400089, Lutherville, Maryland
  - Tufts Medical Center- Site Number : 8400003, Boston, Massachusetts
  - Boston Clinical Trials- Site Number : 8400178, Boston, Massachusetts
  - Neurology Center of New England- Site Number : 8400164, Foxborough, Massachusetts
  - The Elliot Lewis Center- Site Number : 8400033, Wellesley, Massachusetts
  - UMass Memorial Medical Center - University Campus- Site Number : 8400028, Worcester, Massachusetts
  - Henry Ford Hospital- Site Number : 8400091, Detroit, Michigan
  - Michigan Institute for Neurological Disorders- Site Number : 8400004, Farmington Hills, Michigan
  - Trinity Health Grand Rapids- Site Number : 8400150, Grand Rapids, Michigan
  - Memorial Healthcare Institute for Neuroscience- Site Number : 8400123, Owosso, Michigan
  - Rochester Medical Group- Site Number : 8400172, Rochester Hills, Michigan
  - Minneapolis Clinic of Neurology - Golden Valley- Site Number : 8400077, Golden Valley, Minnesota
  - M Health Fairview University of Minnesota Medical Center - East Bank- Site Number : 8400056, Minneapolis, Minnesota
  - Minnesota Center for Multiple Sclerosis- Site Number : 8400073, Plymouth, Minnesota
  - Sharlin Health and Neurology- Site Number : 8400016, Ozark, Missouri
  - Washington University- Site Number : 8400076, St Louis, Missouri
  - Cleveland Clinic Lou Ruvo Center for Brain Health Las Vegas- Site Number : 8400045, Las Vegas, Nevada
  - Renown Regional Medical Center- Site Number : 8400066, Reno, Nevada
  - Dartmouth-Hitchcock Medical Center - Lebanon - 1 Medical Center Drive- Site Number : 8400098, Lebanon, New Hampshire
  - Rutgers University- Site Number : 8400067, New Brunswick, New Jersey
  - Holy Name Medical Center- Site Number : 8400101, Teaneck, New Jersey
  - The University of New Mexico- Site Number : 8400090, Albuquerque, New Mexico
  - Dent Neurologic Institute - Amherst- Site Number : 8400129, Amherst, New York
  - Icahn School of Medicine at Mount Sinai- Site Number : 8400011, New York, New York
  - Columbia University Irving Medical Center- Site Number : 8400088, New York, New York
  - Stony Brook University- Site Number : 8400094, Stony Brook, New York
  - Piedmont HealthCare - Lake Norman Neurology- Site Number : 8400002, Charlotte, North Carolina
  - Raleigh Neurology Associates- Site Number : 8400014, Raleigh, North Carolina
  - Atrium Health - Wake Forest Baptist - Shepherd- Site Number : 8400040, Winston-Salem, North Carolina
  - Sanford Brain and Spine Center- Site Number : 8400085, Fargo, North Dakota
  - Riverhills Neuroscience- Site Number : 8400007, Cincinnati, Ohio
  - University of Cincinnati Medical Center- Site Number : 8400117, Cincinnati, Ohio
  - The Ohio State University- Site Number : 8400009, Columbus, Ohio
  - The Boster Center for Multiple Sclerosis- Site Number : 8400006, Columbus, Ohio
  - UC Health - Elizabeth Place- Site Number : 8400008, Dayton, Ohio
  - Oklahoma Medical Research Foundation- Site Number : 8400039, Oklahoma City, Oklahoma
  - Providence St. Vincent's Medical Center- Site Number : 8400052, Portland, Oregon
  - Penn State Health Milton South Hershey Medical Center- Site Number : 8400176, Hershey, Pennsylvania
  - Thomas Jefferson University Hospital- Site Number : 8400035, Philadelphia, Pennsylvania
  - Premier Neurology- Site Number : 8400047, Greer, South Carolina
  - Hope Neurology- Site Number : 8400019, Knoxville, Tennessee
  - Vanderbilt Multiple Sclerosis Center- Site Number : 8400130, Nashville, Tennessee
  - Neurology Consultants of Dallas - Lyndon B Johnson Freeway- Site Number : 8400152, Dallas, Texas
  - North Texas Institute of Neurology & Headache - Plano- Site Number : 8400083, Plano, Texas
  - Neurology Center of San Antonio- Site Number : 8400099, San Antonio, Texas
  - Texas Institute for Neurological Disorders - Sherman- Site Number : 8400018, Sherman, Texas
  - University of Vermont Medical Center- Site Number : 8400042, Burlington, Vermont
  - Inova Schar Cancer Institute - Fairfax - Innovation Park Drive- Site Number : 8400109, Fairfax, Virginia
  - Riverside Neurology Specialists - Newport News- Site Number : 8400132, Newport News, Virginia
  - Multiple Sclerosis Center of Greater Washington (MSCGW)- Site Number : 8400128, Vienna, Virginia
  - Sentara Family Medicine Physicians - Virginia Beach - Glenn Mitchell Drive- Site Number : 8400168, Virginia Beach, Virginia
  - Swedish Medical Center - Seattle- Site Number : 8400078, Seattle, Washington
  - West Virginia University School of Medicine- Site Number : 8400131, Morgantown, West Virginia
  - Wheaton Franciscan Healthcare - St Francis- Site Number : 8400034, Milwaukee, Wisconsin
  - Medical College of Wisconsin - Milwaukee Campus- Site Number : 8400038, Milwaukee, Wisconsin
- Argentina (5):
  - Investigational Site Number : 0320003, Rosario, Santa Fe Province
  - Investigational Site Number : 0320002, Buenos Aires
  - Investigational Site Number : 0321010, Buenos Aires
  - Investigational Site Number : 0320007, Buenos Aires
  - Investigational Site Number : 0320001, Buenos Aires
- Australia (3):
  - Investigational Site Number : 0360005, Saint Leonards, New South Wales
  - Investigational Site Number : 0360001, Woolloongabba, Queensland
  - Investigational Site Number : 0360002, Melbourne, Victoria
- Belgium (6):
  - Investigational Site Number : 0560001, Bruges
  - Investigational Site Number : 0560008, Brussels
  - Investigational Site Number : 0560006, Ghent
  - Investigational Site Number : 0560007, Kortrijk
  - Investigational Site Number : 0560003, Melsbroek
  - Investigational Site Number : 0560005, Overpelt
- Brazil (15):
  - Centro de Diagnostico e Pesquisa da Osteoporose do Espirito Santo- Site Number : 0760029, Vitória, Espírito Santo
  - Centro de Pesquisas da Clínica IBIS- Site Number : 0760030, Salvador, Estado de Bahia
  - L2IP - Instituto de Pesquisas Clínicas- Site Number : 0760003, Brasília, Federal District
  - Universidade Federal de Goias- Site Number : 0760024, Goiânia, Goiás
  - Freire Pesquisa Clínica - Belo Horizonte - Rua Piauí- Site Number : 0760025, Belo Horizonte, Minas Gerais
  - Instituto de Neurologia de Curitiba - Ecoville- Site Number : 0760001, Curitiba, Paraná
  - Hospital Moinhos de Vento- Site Number : 0760005, Porto Alegre, Rio Grande do Sul
  - IMV Pesquisa Neurológica- Site Number : 0760031, Porto Alegre, Rio Grande do Sul
  - Instituto Ceos- Site Number : 0760028, Porto Alegre, Rio Grande do Sul
  - Clínica Neurológica- Site Number : 0760007, Joinville, Santa Catarina
  - Prognosis Centro de Pesquisa- Site Number : 0760032, Santo André, São Paulo
  - CPHosp Medicina, Ensino e Pesquisa (CPQuali)- Site Number : 0760002, São Paulo
  - PSEG Centro de Pesquisa Clínica- Site Number : 0760021, São Paulo
  - Jordy Sinapse- Site Number : 0760004, São Paulo
  - Hospital Israelita Albert Einstein- Site Number : 0760026, São Paulo
- Bulgaria (9):
  - Investigational Site Number : 1000009, Blagoevgrad
  - Investigational Site Number : 1000008, Panagyurishte
  - Investigational Site Number : 1000007, Pazardzhik
  - Investigational Site Number : 1000002, Pleven
  - Investigational Site Number : 1000010, Pleven
  - Investigational Site Number : 1000004, Sofia
  - Investigational Site Number : 1000001, Sofia
  - Investigational Site Number : 1000006, Sofia
  - Investigational Site Number : 1000005, Sofia
- Canada (14):
  - Investigational Site Number : 1240011, Calgary, Alberta
  - Investigational Site Number : 1240005, Burnaby, British Columbia
  - Investigational Site Number : 1240010, Vancouver, British Columbia
  - Investigational Site Number: 1240018, Moncton, New Brunswick
  - Investigational Site Number : 1240014, London, Ontario
  - Investigational Site Number : 1240002, Ottawa, Ontario
  - Investigational Site Number : 1240015, Toronto, Ontario
  - Investigational Site Number : 1240012, Toronto, Ontario
  - Investigational Site Number : 1240001, Gatineau, Quebec
  - Investigational Site Number : 1240008, Lévis, Quebec
  - Investigational Site Number : 1240009, Montreal, Quebec
  - Investigational Site Number : 1240016, Pointe-Claire, Quebec
  - Investigational Site Number : 1240003, Québec, Quebec
  - Investigational Site Number : 1240006, Sherbrooke, Quebec
- Chile (3):
  - Investigational Site Number : 1520003, Las Condes, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520002, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520001, Santiago, Reg Metropolitana de Santiago
- China (16):
  - Investigational Site Number : 1560007, Beijing
  - Investigational Site Number : 1560005, Beijing
  - Investigational Site Number : 1560008, Beijing
  - Investigational Site Number : 1560003, Changchun
  - Investigational Site Number : 1560011, Changsha
  - Investigational Site Number : 1560004, Chengdu
  - Investigational Site Number : 1560045, Fuzhou
  - Investigational Site Number : 1560002, Guangzhou
  - Investigational Site Number : 1561027, Harbin
  - Investigational Site Number : 1560010, Jiazhuang
  - Investigational Site Number : 1560001, Shanghai
  - Investigational Site Number : 1560006, Taiyuan
  - Investigational Site Number : 1560012, Tianjin
  - Investigational Site Number : 1560009, Wuhan
  - Investigational Site Number : 1560013, Xi'an
  - Investigational Site Number : 1560034, Zhengzhou
- Czechia (8):
  - Investigational Site Number : 2030011, Brno
  - Investigational Site Number : 2030005, Brno
  - Investigational Site Number : 2030002, Hradec Králové
  - Investigational Site Number : 2030006, Jihlava
  - Investigational Site Number : 2030007, Ostrava
  - Investigational Site Number : 2030008, Prague
  - Investigational Site Number : 2030009, Teplice
  - Investigational Site Number : 2030001, Zlín
- France (14):
  - Investigational Site Number : 2500011, Bron
  - Investigational Site Number : 2500005, Créteil
  - Investigational Site Number : 2500017, Gonesse
  - Investigational Site Number : 2500006, La Tronche
  - Investigational Site Number : 2500009, Lille
  - Investigational Site Number : 2500015, Montpellier
  - Investigational Site Number : 2500016, Nancy
  - Investigational Site Number : 2500002, Nice
  - Investigational Site Number : 2500018, Orsay
  - Investigational Site Number : 2500007, Paris
  - Investigational Site Number : 2500014, Paris
  - Investigational Site Number : 2500003, Rennes
  - Investigational Site Number : 2500010, Saint-Herblain
  - Investigational Site Number : 2500001, Strasbourg
- Germany (11):
  - Investigational Site Number : 2760009, Bielefeld
  - Investigational Site Number : 2760010, Bochum
  - Investigational Site Number : 2760012, Dresden
  - Investigational Site Number : 2760002, Düsseldorf
  - Investigational Site Number : 2760013, Erbach im Odenwald
  - Investigational Site Number : 2760014, Heidelberg
  - Investigational Site Number : 2760007, Jena
  - Investigational Site Number : 2760003, Leipzig
  - Investigational Site Number : 2760008, Marburg
  - Investigational Site Number : 2760006, Münster
  - Investigational Site Number : 2760001, Ulm
- Greece (5):
  - Investigational Site Number : 3000003, Athens
  - Investigational Site Number : 3000005, Athens
  - Investigational Site Number : 3000004, Ioannina
  - Investigational Site Number : 3000001, Larissa
  - Investigational Site Number : 3000002, Thessaloniki
- Hungary (4):
  - Investigational Site Number : 3480003, Budapest
  - Investigational Site Number : 3480004, Budapest
  - Investigational Site Number : 3480006, Budapest
  - Investigational Site Number : 3480002, Győr
- India (4):
  - Investigational Site Number : 3560024, Bengaluru
  - Investigational Site Number : 3560008, Hyderabad
  - Investigational Site Number : 3560017, New Delhi
  - Investigational Site Number : 3560006, Shimla
- Italy (23):
  - Investigational Site Number : 3800034, Augusta, Catania
  - Investigational Site Number : 3800025, Cona, Ferrara
  - Investigational Site Number : 3800004, Florence, Firenze
  - Investigational Site Number : 3800011, Genoa, Genova
  - Investigational Site Number : 3800008, Pozzilli, Isernia
  - Investigational Site Number : 3800002, Milan, Milano
  - Investigational Site Number : 3800016, Milan, Milano
  - Investigational Site Number : 3800010, Naples, Napoli
  - Investigational Site Number : 3800006, Cefalù, Palermo
  - Investigational Site Number : 3800015, Rome, Roma
  - Investigational Site Number : 3800001, Rome, Roma
  - Investigational Site Number : 3800013, Rome, Roma
  - Investigational Site Number : 3800021, Rome, Roma
  - Investigational Site Number : 3800035, Gallarate, Varese
  - Investigational Site Number : 3800009, Bologna
  - Investigational Site Number : 3800014, Chieti
  - Investigational Site Number : 3800019, Foggia
  - Investigational Site Number : 3800026, Novara
  - Investigational Site Number : 3800017, Palermo
  - Investigational Site Number : 3800029, Parma
  - Investigational Site Number : 3800005, Pavia
  - Investigational Site Number : 3800003, Perugia
  - Investigational Site Number : 3800030, Ravenna
- Japan (11):
  - Investigational Site Number : 3920003, Kōriyama, Fukushima
  - Investigational Site Number : 3920014, Asahikawa, Hokkaido
  - Investigational Site Number : 3920007, Himeji, Hyōgo
  - Investigational Site Number : 3920010, Sagamihara, Kanagawa
  - Investigational Site Number : 3920015, Higashi-Matsuyama, Saitama
  - Investigational Site Number : 3920016, Kodaira, Tokyo
  - Investigational Site Number : 3920002, Chiba
  - Investigational Site Number : 3920013, Fukuoka
  - Investigational Site Number : 3920001, Kyoto
  - Investigational Site Number : 3920011, Tokyo
  - Investigational Site Number : 3920012, Tokyo
- Investigational Site Number : 5280002, Rotterdam, Netherlands
- Poland (9):
  - Investigational Site Number : 6160002, Plewiska, Greater Poland Voivodeship
  - Investigational Site Number : 6160012, Poznan, Greater Poland Voivodeship
  - Investigational Site Number : 6160018, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Investigational Site Number : 6160005, Krakow, Lesser Poland Voivodeship
  - Investigational Site Number : 6160006, Rzeszów, Podkarpackie Voivodeship
  - Investigational Site Number : 6160007, Bialystok, Podlaskie Voivodeship
  - Investigational Site Number : 6160010, Katowice, Silesian Voivodeship
  - Investigational Site Number : 6160011, Katowice, Silesian Voivodeship
  - Investigational Site Number : 6160004, Zabrze, Silesian Voivodeship
- Portugal (5):
  - Investigational Site Number : 6200001, Braga
  - Investigational Site Number : 6200011, Lisbon
  - Investigational Site Number : 6200007, Lisbon
  - Investigational Site Number : 6200006, Lisbon
  - Investigational Site Number : 6200002, Matosinhos Municipality
- Investigational Site Number : 6820001, Riyadh, Saudi Arabia
- South Korea (5):
  - Investigational Site Number : 4100001, Goyang-si, Gyeonggi-do
  - Investigational Site Number : 4100007, Seongnam-si, Gyeonggi-do
  - Investigational Site Number : 4100002, Seoul, Seoul-teukbyeolsi
  - Investigational Site Number : 4100004, Seoul, Seoul-teukbyeolsi
  - Investigational Site Number : 4100003, Seoul, Seoul-teukbyeolsi
- Spain (22):
  - Investigational Site Number : 7240018, Murcia, Almería
  - Investigational Site Number : 7240016, Barcelona, Barcelona [Barcelona]
  - Investigational Site Number : 7240010, Barcelona, Barcelona [Barcelona]
  - Investigational Site Number : 7240009, Barakaldo, Basque Country
  - Investigational Site Number : 7240011, L'Hospitalet de Llobregat, Catalunya [Cataluña]
  - Investigational Site Number : 7240012, Donostia / San Sebastian, Gipuzkoa
  - Investigational Site Number : 7240024, Girona, Girona [Gerona]
  - Investigational Site Number : 7240013, Las Palmas de Gran Canaria, Las Palmas
  - Investigational Site Number : 7240015, Lleida, Lleida [Lérida]
  - Investigational Site Number : 7240017, Majadahonda, Madrid
  - Investigational Site Number : 7240001, Pozuelo de Alarcón, Madrid
  - Investigational Site Number : 7240014, Pontevedra, Pontevedra [Pontevedra]
  - Investigational Site Number : 7240007, Seville, Sevilla
  - Investigational Site Number : 7240004, Córdoba
  - Investigational Site Number : 7240006, Madrid
  - Investigational Site Number : 7240023, Madrid
  - Investigational Site Number : 7240002, Madrid
  - Investigational Site Number : 7240003, Madrid
  - Investigational Site Number : 7240022, Madrid
  - Investigational Site Number : 7240005, Málaga
  - Investigational Site Number : 7240008, Valencia
  - Investigational Site Number : 7240025, Zaragoza
- Sweden (4):
  - Investigational Site Number : 7520001, Gothenburg
  - Investigational Site Number : 7520005, Huddinge
  - Investigational Site Number : 7520003, Malmo
  - Investigational Site Number : 7520002, Stockholm
- Turkey (Türkiye) (19):
  - Investigational Site Number : 7920018, Ankara
  - Investigational Site Number : 7920011, Ankara
  - Investigational Site Number : 7920020, Bursa
  - Investigational Site Number : 7920013, Bursa
  - Investigational Site Number : 7920005, Eskişehir
  - Investigational Site Number : 7920012, Istanbul
  - Investigational Site Number : 7920002, Istanbul
  - Investigational Site Number : 7920016, Istanbul
  - Investigational Site Number : 7920009, Istanbul
  - Investigational Site Number : 7920007, Istanbul
  - Investigational Site Number : 7920019, Izmir
  - Investigational Site Number : 7920008, Izmir
  - Investigational Site Number : 7920001, İzmit
  - Investigational Site Number : 7920014, Kayseri
  - Investigational Site Number : 7920015, Konya
  - Investigational Site Number : 7920006, Mersin
  - Investigational Site Number : 7920004, Samsun
  - Investigational Site Number : 7920003, Sultangazi
  - Investigational Site Number : 7920017, Van
- Ukraine (8):
  - Investigational Site Number : 8040001, Chernivtsi
  - Investigational Site Number : 8040009, Ivano-Frankivsk
  - Investigational Site Number : 8040003, Ivano-Frankivsk
  - Investigational Site Number : 8040006, Kyiv
  - Investigational Site Number : 8040008, Lutsk
  - Investigational Site Number : 8040004, Lviv
  - Investigational Site Number : 8040002, Lviv
  - Investigational Site Number : 8040005, Vinnytsia
- United Kingdom (11):
  - Investigational Site Number : 8260011, Gwent, Blaenau Gwent
  - Investigational Site Number : 8260001, Exeter, Devon
  - Investigational Site Number : 8260013, London, England
  - Investigational Site Number : 8260006, Newcastle upon Tyne, England
  - Investigational Site Number : 8260010, Inverness, Highland
  - Investigational Site Number : 8260003, Canterbury, Kent
  - Investigational Site Number : 8260008, Salford, Manchester
  - Investigational Site Number : 8260004, Oxford, Oxfordshire
  - Investigational Site Number : 8260005, Swansea, Swansea [Abertawe Gb-ata]
  - Investigational Site Number : 8260007, Cardiff, Vale of Glamorgan, the
  - Investigational Site Number : 8260009, Liverpool

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: Multiple Sclerosis Website — https://www.sanofistudies.com/JQ2Z/
- See also: EFC17504 Plain Language Results Summary — https://sanofi.trialsummaries.com/Study/StudyDetails?id=25596&tenant=MT_SNY_9011